CLINICAL TRIAL: NCT01721720
Title: The Neurobehavioral, Environmental and Genetic Factors Impacting the Clinical Course of Attention Deficit Hyperactivity Disorder
Brief Title: Genetic, Brain Structure, and Environmental Effects on ADHD
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120202; 12-HG-0202
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Peer and Family Networks; Longitudinal Outcome; MRI Imaging; Genetics; Childhood Psychiatric Disorders; Natural History
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with and without ADHD: Participants with and without ADHD

SUMMARY:
Background:

- Attention deficit hyperactivity disorder (ADHD) is one of the most common and inheritable of all neuropsychiatric disorders. It causes problems with attention and impulse control. However, the genetic component of ADHD has not been fully studied, including how genes interact with the environment. Researchers want to study children and adults who have ADHD. They will look at how genetic, brain structure, and environmental factors affect ADHD in children and adults.

Objectives:

- To study genetic, brain structure, and environmental factors in ADHD in children and adults.

Eligibility:

- Individuals at least 3 years of age who have ADHD.

Design:

* Participants will be screened with a physical exam and medical history.
* Participants will be interviewed about their ADHD. They will also complete behavior and psychological tests. Parents or guardians will complete the tests along with participants under 18 years of age.
* Participants will provide saliva or blood samples.
* Participants will also have imaging studies of the brain.
* Participants under 25 years of age will return once a year to repeat the tests. Those over 25 years of age will have only the one set of tests. Those who are starting stimulant drugs and who are receiving behavioral treatment for the first time will also have another set of tests 12 weeks after the start of treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

This study aims to provide novel phenotypes for genomic studies into Attention- Deficit Hyperactivity Disorder (ADHD), one of the most common and heritable of all neuropsychiatric disorders. It proposes to split the disorder into neurobiologically more meaningful entities by delineating subgroups based on neurobehavioral profiles. It will also explore factors that impact clinical course, focusing on the neural effects of treatment and the role of the child s social environment.

POPULATION AND DESIGN:

Using a prospective longitudinal design, a group of children and adolescents with ADHD will be followed. Additionally, families that have several members affected by ADHD will be recruited.

OUTCOMES:

The study will link the onset and clinical course of ADHD with genotype, brain structure and function, behavior and the child s social environment.

ELIGIBILITY:
* INCLUSION CRITERIA FOR ALL PARTICIPANTS:

Three or more years of age with no upper limit for age at time of enrollment. The lower limit of 3 years of age is chosen as it is difficult to diagnose ADHD below this age, but the diagnosis can be reliably made from age 3 onwards. As this study examines the developmental trajectories of ADHD into adulthood, no upper age limit has been set.

INCLUSION CRITERIA FOR CLINICAL POPULATIONS:

Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) defined ADHD. The DSM-IV diagnosis of ADHD will be based on the Parent Diagnostic Interview for Children and Adolescents in participants 18 years or age and younger and the

Structured clinical interview for the Diagnosis of DSM Disorders for participants above 18 years of age. We include all forms of ADHD in DSM-5 (i.e. combined, predominately hyperactive/impulsive, predominately inattentive and other specified presentations). ADHD is rarely found in isolation and comorbidity is common. Thus the protocol will include individuals with ADHD and the

following disorders: oppositional defiant disorder, conduct disorder, anxiety disorders (generalized anxiety, specific phobias), tic disorders, mood disorders (dysthymia, depression); specific learning disabilities and disruptive mood dysregulation disorder.

We will also include families where there is a incidence of >30% of ADHD in first, second and third degree relatives. This level is chosen as it is well above the incidence rate of ADHD in the general population (~5-7%). Additional inclusion criteria are families where the proband has at least one sibling and only one or neither parent is affected.

In studying the acute effects of treatment we will include all participants with ADHD who are starting psychostimulant medications for the first time (all psychostimulant preparations are included). We will also include participants with ADHD who are receiving behavioral

management for ADHD for the first time.

INCLUSIONS CRITERIA FOR THE FAMILY STUDY:

We will also include families where there is a incidence of >30% of ADHD in first, second and third degree relatives. This level is chosen as it is well above the incidence rate of ADHD in the general population (~5-7%). Additional inclusion criteria are families where the proband has at least one sibling and only one or neither parent is affected.

We have already identified families of our currently enrolled probands in which at least 4 other first, second or third degree relatives have a current diagnosis of ADHD or had this diagnosis in childhood (and have a similar number of unaffected relatives). We will recruit further families with a similar density of individual affected by ADHD.

EXCLUSION CRITERIA FOR ALL PARTICIPANTS:

Full scale IQ of less than 70. Below this level a child is considered to have global intellectual disability (classified in DSM-IVR as mental retardation). By definition this means the individual cannot be considered to be a healthy control . While many individual with IQ below 70 have symptoms of ADHD, the diagnosis is complicated by problems in assessing attentional abilities.

Finally, there are often issues around the ability to give informed consent in adults with global intellectual disability.

Birth before 32 weeks of gestation. Premature birth can have a profound effect on brain function and structure.

Presence or history of medical conditions known to affect cerebral anatomy (eg epilepsy, history of stroke). Genetic syndromes which are associated with well-established alterations of gross cerebral structure- such as NF1, tuberous sclerosis and some forms of epilepsy. Children with known microdeletion syndromes will not be excluded provided (1) the syndrome is not known to be associated with alteration of cerebral anatomy (detectable on current clinical MRI sequences) and (2) other exclusionary criteria do not apply such as global intellectual impairment (defined in this protocol as IQ above 70). Data from these individuals with microdeletion syndromes will

not however be included in GWAS due to analytic complications.

Dental braces (as these distort the MRI image). Metal in the body or other contraindications for MRI scanning. For females who have reached menarche and have not yet past menopause: pregnancy or inability or unwillingness to undergo pregnancy testing (for MRI

safety).

For participants 60 years or older. Folstein mini mental state examination score of 26 or greater. This is a widely accepted screening test for dementia.

ADDITIONAL EXCLUSION CRITERIA FOR HEALTHY VOLUNTEERS ONLY: Presence of any DSM-IV psychiatric disorder in the subject or current use of psychiatric medication.

ADDITIONAL EXCLUSION CRITERIA FOR THE CLINICAL POPULATION ONLY:

Some neuropsychiatric disorders are either so rare or associated with such profound alterations of brains structure and function that they will be excluded. This includes psychotic disorders (including schizophrenia, psychosis NOS) bipolar affective disorder; autism, substance dependence; dementia.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children, adolescents, and adults with Attention Deficit Hyperactivity Disorder and healthy controls. Some participants will be from families that have many individuals affected by ADHD.
Sampling Method: Non-Probability Sample
Enrollment: 1091 (Actual)
Dates: Start 2012-11-09 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Brain MRI | yearly or at the participant's availability
  Trajectories of brain development

SECONDARY OUTCOMES:
DNA collection, clinical interviews, social network information gathering | yearly or at the participant's convenience
  To explore the neural, genomic and socio-environmental factors that determine the course of ADHD

CONTACTS AND LOCATIONS:
Overall Officials: Wallace P Shaw, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified medical information will be placed in a NIH repository (e.g., Biomedical Translational Research Information System (BTRIS)) in accordance to NIH policies. We will also share genomic and phenotypic data in controlled access databases such as dbGAP (database of Genotypes and Phenotypes). Other databases may be used as approved by NIH for the sharing of de-identified data.
Supporting Information: Study Protocol
Time Frame: The timeline for data sharing will follow the NHGRI Genomic Data Sharing Policy. Currently data is deposited following IRB review once the study data collection is complete and the data has undergone quality control steps.
Access Criteria: Access requests for specific research purposes using NIH controlled-access data are reviewed by NIH Data Access Committees (DACs).

REFERENCES:
- [Derived] Sudre G, Norman L, Bouyssi-Kobar M, Price J, Shastri GG, Shaw P. A Mega-analytic Study of White Matter Microstructural Differences Across 5 Cohorts of Youths With Attention-Deficit/Hyperactivity Disorder. Biol Psychiatry. 2023 Jul 1;94(1):18-28. doi: 10.1016/j.biopsych.2022.09.021. Epub 2022 Sep 26. PMID 36609028
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-HG-0202.html